CLINICAL TRIAL: NCT02728557
Title: The Roles of the Therapeutic Alliance in Understanding the Effects of Attachment Orientations on Outcome in Psychotherapy
Brief Title: Supportive and Supportive-Expressive Treatment for Depression
Acronym: SSETD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Sigal Zilcha Mano, Full Professor, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISF 186.15
Record Dates: First submitted 2016-03-15; First posted 2016-04-05 (Estimated); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder
Keywords: Therapeutic alliance; Psychotherapy; Psychodynamic psychotherapy; supportive-expressive treatment; Process research; Attachment theory; Attachment orientation; Mechanism of change in psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive psychotherapy (Experimental): Participants will receive supportive therapy.
  Interventions: Behavioral: Supportive Therapy
- Supportive-expressive psychotherapy (Experimental): Participants will receive supportive-expressive therapy.
  Interventions: Behavioral: Supportive-Expressive Therapy

INTERVENTIONS:
Behavioral: Supportive-Expressive Therapy — Supportive-expressive psychotherapy for depressive disorder for 16 weeks.
  Arms: Supportive-expressive psychotherapy
Behavioral: Supportive Therapy — Supportive psychotherapy for depressive disorder for 16 weeks.
  Arms: Supportive psychotherapy

SUMMARY:
This study will assign patients to two types of psychotherapies in treating people with a major depression disorder, expressive versus supportive techniques, and will examine their ability to benefit from treatment based on their attachment orientation. This is a four month protocol, with a year follow up period, will compare patients receiving supportive-expressive treatment with either expressive focus or supportive focus.

DETAILED DESCRIPTION:
One hundred patients suffering from major depression will participate in 16 sessions of supportive-expressive treatment. Patients will be randomized to one of two conditions: one that places a greater emphasis on supportive techniques, or one that places a greater emphasis on expressive techniques. These two conditions (supportive vs. expressive) hold the potential of either complementing or counter-complementing patients' attachment orientations (e.g., for a patient with higher levels of attachment anxiety, the supportive condition is complementary while the expressive is counter-complementary; the reverse is true for a patient with higher levels of attachment avoidance). Importantly, this study will employ multiple complementary methods, which will include session-by-session self-report alliance questionnaires from both patient and therapist, as well as a cognitive task assessing patients' relationship expectations, and behavioral observations of therapist-patient interactions. This study will be the first to utilize such a combination of methodologies in psychotherapy research and the first to examine the proposed mediation model. It will also be the first to manipulate the use of techniques in order to experimentally examine whether therapeutic techniques can be utilized to develop more efficient treatment models, based on the two transdiagnostic concepts of attachment and alliance. The findings will contribute both to our understanding of the relevance of attachment theory to psychotherapy research, and to the growing empirical literature on targeting transdiagnostic concepts (here, attachment and alliance) that cut across many disorders and treatment orientations. These transdiagnostic concepts can be utilized in the move towards tailoring existing psychological interventions to specific individuals according to their attachment orientations.

ELIGIBILITY:
Inclusion Criteria:

* Meeting MDD diagnostic criteria using the structured clinical interviews for DSM-V and scoring more than 14 on the 17-item Hamilton rating scale for depression at two evaluations (one week apart).
* If on medication, patients' dosage must be stable for at least three months prior to entering the study, and they must be willing to maintain stable dosage for the duration of treatment
* Age between 18 and 60
* Hebrew language fluency
* Provision of written informed consent.

Exclusion Criteria:

* Current risk of suicide or self-harm
* Current substance abuse disorders
* Current or past schizophrenia or psychosis, bipolar disorder, or severe eating disorder requiring medical monitoring
* History of organic mental disease
* Currently in psychotherapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2023-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sigal Zilcha Mano, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Mount Carmel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacol Bull. 1993;29(2):321-6. PMID 8290681
- [Background] Horowitz LM, Rosenberg SE, Baer BA, Ureno G, Villasenor VS. Inventory of interpersonal problems: psychometric properties and clinical applications. J Consult Clin Psychol. 1988 Dec;56(6):885-92. doi: 10.1037//0022-006x.56.6.885. No abstract available. PMID 3204198
- [Derived] Zilcha-Mano S, Webb CA. Identifying who benefits most from supportive versus expressive techniques in psychotherapy for depression: Moderators of within- versus between-individual effects. J Consult Clin Psychol. 2024 Mar;92(3):187-197. doi: 10.1037/ccp0000868. Epub 2023 Dec 7. PMID 38059944
- [Derived] Zilcha-Mano S, Ben David-Sela T. Is alliance therapeutic in itself? It depends. J Couns Psychol. 2022 Nov;69(6):786-793. doi: 10.1037/cou0000627. Epub 2022 Aug 4. PMID 35925745
- [Derived] Zilcha-Mano S, Dolev-Amit T, Fisher H, Ein-Dor T, Strauss B. Patients' individual differences in implicit and explicit expectations from the therapist as a function of attachment orientation. J Couns Psychol. 2021 Nov;68(6):682-695. doi: 10.1037/cou0000503. Epub 2021 Jun 28. PMID 34180691
- [Derived] Zilcha-Mano S, Dolev T, Leibovich L, Barber JP. Identifying the most suitable treatment for depression based on patients' attachment: study protocol for a randomized controlled trial of supportive-expressive vs. supportive treatments. BMC Psychiatry. 2018 Nov 12;18(1):362. doi: 10.1186/s12888-018-1934-1. PMID 30419875

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive-expressive Psychotherapy | Supportive Psychotherapy
Started | 50 | 50
Completed | 48 | 45
Not Completed | 2 | 5
Not completed — Dissatisfaction with assigned treatment | 1 | 3
Not completed — Dissatisfaction with research tasks | 0 | 1
Not completed — Scheduling or change in availability | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supportive Psychotherapy | Supportive-expressive Psychotherapy | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.02 (6.9) | 31.5 (9.6) | 31.2 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 21 | 22 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 50 | 50 | 100
HRSD [Mean (Standard Deviation); unit: Unit on a scale] — Hamilton Rating Scale for Depression
  Unit on a scale | 20.84 (3.588) | 21.00 (3.881) | 20.92 (3.719)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HRSD)
Description: A clinically administered measure assessing the severity of depression.
  The Hamilton is the standard measure of depression severity for clinical trials.
  The scoring is based on the first 17-items of the Hamilton.
  0-7 = NORMAL 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression >=23 = Very Severe Depression
  Hamilton Rating Scale for Depression, developed by Max Hamilton in 1967, is a widely used tool for assessing the severity of depression in adults.
  17 items covering various aspects of depression experienced in the past week. Each item is rated on a 3-point or 5-point scale depending on the specific symptom.
  Total score (sum score) provides an indication of depression severity.
  The range is 0-52
Time Frame: Slope from baseline to week 16.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supportive-expressive Psychotherapy | Supportive Psychotherapy
Number analyzed (Participants) | 50 | 50
units on a scale
  Change from baseline to week 16 | 12.32 (6.52) | 12.06 (6.26)
  Baseline | 20.20 (4.106) | 20.08 (3.702)
Statistical Analysis 1: Comparison: Supportive-expressive Psychotherapy vs Supportive Psychotherapy; A model with two three-way interactions of time by treatment condition by attachment orientation (Time Å~ Treatment condition Å~ Attachment anxiety, Time Å~ Treatment condition Å~ Attachment avoidance) along the lower-level effects to predict differences in the slope of change in outcome. The threshold for statistical significance was p>0.05; Test type: Other — MLM models; p = .016, MLM; MLM

2. Secondary Outcome: Beck Depression Inventory (BDI)
Description: Beck Depression Inventory; measuring depression by a self-report measure; higher means worse outcomes.
  The Beck Depression Inventory consists of 21 multiple-choice questions. Each question presents different statements reflecting varying intensities of a particular depressive symptom.
  Each question has scores ranging from 0 (no symptoms) to 3 (most severe symptoms).
  The total score is obtained by summing up the scores of all chosen responses.
  Based on the total score, there are different interpretations of depression severity:
  Scores in the 0-13 range suggest minimal or no depression. Scores between 14-19 indicate mild depression. Scores from 20-28 reflect moderate depression. Scores 29 and above suggest severe depression. Range 0-63
Time Frame: Slope from baseline to week 16. Measured at baseline, every week for 16 weeks of treatment, then once a month for four months and follow up after a year; Scores are provided for baseline and change from baseline to week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supportive-expressive Psychotherapy | Supportive Psychotherapy
Number analyzed (Participants) | 50 | 50
units on a scale
  Change from baseline to week 16 | 16.62 (9.63) | 13.36 (10.59)
  Baseline | 27.55 (8.617) | 25.76 (7.604)

3. Secondary Outcome: Outcome Questionnaire (OQ)
Description: Outcome Questionnaire; measuring Symptom Distress, Interpersonal Relationships, Social Role; higher levels mean worse outcome.
  Outcome Questionnaire-30 (OQ-30; Lambert et al., 1996). OQ-30 is a 30-item self-report measure assessing distress, designed to measure patient progress.
  Items were rated on a 5 point likert scale ranging from 0 (never) to 4 (almost always). The OQ-30 has three subscales assessing symptom distress, interpersonal relations, and social role performance.
  A total score is calculated by sum scores. Range 0-120
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supportive-expressive Psychotherapy | Supportive Psychotherapy
Number analyzed (Participants) | 50 | 50
units on a scale
  Changes from baseline to week 16 | 32.26 (20.54) | 26.33 (18.44)
  Baseline | 73.435 (13.504) | 69.519 (13.213)

4. Other Pre Specified Outcome: Inventory of Interpersonal Problems Circumplex (IIP-C)
Description: Inventory of Interpersonal Problems Circumplex; measuring interpersonal problems; higher means worse outcomes Inventory of Interpersonal Problems-Circumplex (IIP-C). The IIP-C is a 32-item self-report questionnaire assessing interpersonal difficulties and distress.
  Patients rate two types of items: interpersonal behaviors that are "hard for you to do" (e.g., "it is hard for me to let other people know when I am angry") and interpersonal behaviors that "you do too much" (e.g., "I am too afraid of other people").
  Ratings of the degree to which each problem is distressing are made on a 5-point scale, ranging from 0 (not at all) to 4 (extremely).
  Calculated as a sum score. Range 0 -128
Time Frame: Measured at baseline, six times during the treatment (weeks 1, 2, 4, 8, 12, 16), then once a month for four months and follow up after a year; reports refer to baseline and changes from baseline to week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supportive-expressive Psychotherapy | Supportive Psychotherapy
Number analyzed (Participants) | 50 | 50
units on a scale
  Changes from baseline to week 16 | 13.38 (15.92) | 11.94 (12.7)
  Baseline | 55.58 (12.52) | 59.32 (15.306)

5. Other Pre Specified Outcome: Experiences in Close Relationships Questionnaire (ECR)
Description: Experiences in Close Relationships Questionnaire; The measurement data will be aggregated into two sub-scales: anxiety and avoidance; higher scores mean worse outcomes (less secure attachment) Experience in Close Relationships Scale (ECR; Brennan et al., 1998). 36-item self-reported measure. Participants rated the extent to which each item was descriptive of their experiences in close relationships on a 7-point Likert scale ranging from 1 (not at all) to 7 (very much).
  18 items assessed attachment anxiety (e.g., "I worry about being abandoned"). 18 assessed attachment avoidance (e.g., "I prefer not to show a partner how I feel deep down"). The reliability and validity of these scales have been repeatedly demonstrated (Brennan et al., 1998; Mikulincer & Shaver, 2007).
  The score for each subscale is calculated as the average value Range 1-7
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supportive-expressive Psychotherapy | Supportive Psychotherapy
Number analyzed (Participants) | 50 | 50
units on a scale
  Anxiety - change from baseline to week 16 | 0.9 (1.16) | 0.6 (0.97)
  Avoidance - change from baseline to week 16 | 0.54 (0.87) | 0.21 (0.79)
  Anxiety - baseline | 4.07 (1.207) | 4.101 (1.02)
  Avoidance - baseline | 4.202 (1.045) | 4.036 (1.011)

6. Other Pre Specified Outcome: Quality of Life Enjoyment and Satisfaction- Short Version (Q-LES-Q)
Description: Quality of Life Enjoyment and Satisfaction- Short Version; measuring quality of life; higher scores mean better outcomes.
  The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q). It's a self-report measure, meaning the person being assessed completes the questionnaire themselves.
  Purpose: It gauges the degree of enjoyment and satisfaction a person experiences in different areas of their daily functioning.
  Utilize a 5-point Likert scale, ranging from 1 (very poor) to 5 (very good). Higher scores mean better outcomes. Range 1-5. Average score
Time Frame: Measured at baseline, six times during the treatment (weeks 1, 2, 4, 8, 12, 16), then once a month for four months and follow up after a year; reports refer to baseline and change from baseline to week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supportive-expressive Psychotherapy | Supportive Psychotherapy
Number analyzed (Participants) | 50 | 50
units on a scale
  Change from baseline to week 16 | 0.70 (0.73) | 0.48 (0.63)
  Baseline | 2.848 (0.542) | 2.801 (0.505)

ADVERSE EVENTS:
Time Frame: Active phase - baseline to week 16, and then 2 years
Arm/Group | Supportive-expressive Psychotherapy | Supportive Psychotherapy
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Because of COVID, 13 patients were treated remotely. The total number of patients was according to the pre-registration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT02728557/Prot_SAP_000.pdf